CLINICAL TRIAL: NCT01433289
Title: Placebo-Controlled, Dose-Blinded, Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Polyphenon E (EGCG) 14 Day Monotherapy in Antiretroviral Naïve and Experienced, HIV-1-Infected Subjects
Brief Title: Study to Evaluate Safety and Toxicity of Polyphenon E (EGCG) in HIV-1-Infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Filiz Seeborg, Associate Professor Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-21490; R21AT004673 (NIH)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: HIV Infection
Keywords: HIV; safety; toxicity; pharmacokinetics; Polyphenon E; EGCG; green tea; CD4; viral load
MeSH Terms: conditions — HIV Infections | interventions — polyphenon E; epigallocatechin gallate; Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Polyphenon E 1600 mg/day (Experimental): Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Four capsules twice a day.
  Interventions: Drug: Polyphenon E
- Polyphenon E 2400 mg/day (Experimental): Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Six capsules twice a day.
  Interventions: Drug: Polyphenon E
- Polyphenon E 3200 mg/day (Experimental): Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Eight capsules twice a day.
  Interventions: Drug: Polyphenon E
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyphenon E — There will be 3 dose levels and for each dose level, there will be 6 subjects who will receive the study drug and 2 subjects who will be randomized to take placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding dose level will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each dose level is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
  Other Names: EGCG; epigallocatechin gallate; green tea catechin; green tea extract
  Arms: Polyphenon E 1600 mg/day; Polyphenon E 2400 mg/day; Polyphenon E 3200 mg/day
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, toxicity, dosing, and antiviral effects of epigallocatechin gallate (EGCG) in capsule form (Polyphenon® E), administered orally twice daily at three different doses in HIV-1-infected clinically stable, treatment-naïve and treatment-experienced adults not on concomitant antiretroviral (ARV) therapy.

DETAILED DESCRIPTION:
HIV-1 infection ultimately results in impaired specific immune function by virtue of the initial binding of the HIV-1 virion envelope glycoprotein 120 (gp120) to the CD4 receptor in complex with a chemokine receptor on the T-cell surface1. Even though gp120 elicits virus-neutralizing antibodies, HIV-1 eludes the immune system and leads to the onset of AIDS. Ever since the discovery of the virus as the causative agent, there has been an intense effort to develop therapeutic methods to inhibit or prevent infection.2-4 CD4, a cell surface glycoprotein expressed on T cells, plays an important role in the recognition of antigens by T cells and in their activation.5 It also acts as a receptor for HIV-1 as gp120 binds to it via its D1 domain and, uses this interaction to infect CD4+ T cells.5 Therefore, there has been interest in finding molecules that block the binding of gp120 to CD4 (entry inhibitors) as a way of reducing HIV-1 infectivity.

Studies have demonstrated evidence of high affinity binding of EGCG to the CD4 molecule with a Kd of 10nM with subsequent inhibition of gp120 binding to human CD4+ T cells. EGCG binds in the same molecular pocket on CD4, as does HIV-1-gp120 at physiologically relevant concentrations.

This is a phase I, placebo-controlled, dose-blinded, randomized study of Polyphenon® E as monotherapy in participants who are HIV-1-infected with a CD+ T lymphocyte count of at least 250 cells/mm3 and are ARV-naïve or ARV-experienced. There will be 3 dose levels and for each dose level, there will be 6 subjects who will receive the study drug and 2 subjects who will be randomized to take placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding dose level will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each dose level is completed. If at least 4 subjects on the active drug in each dose level have evaluable PK data, subjects will not be replaced. As the inability to achieve adequate EGCG concentrations that are necessary to inhibit HIV-1 replication is a major concern in this study, it is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each dose level. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject. If only a few samples cannot be used (this depends on the individual subject's pharmacokinetic profile, although one or two unevaluable samples will not likely cause a subject's data to be unevaluable), PK analyses can still be performed and will not require subjects to be deemed unevaluable and replaced.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individual as having at least two of the following in any combination obtained from 2 different samples: Positive HIV rapid test or ELISA and Western Blot; HIV RNA PCR>10,000 copies/ml; positive HIV DNA PCR; neutralizable HIV p 24 antigen
* Asymptomatic HIV-1 infected individuals who are either antiretroviral-naive or treatment-experienced. Subjects must have not been on ARV treatment for at least 12 weeks prior to enrollment and not have plans to start ARV treatment within 8 weeks of study initiation.
* Male or female 18 to 65 years of age. Males must use barrier methods of contraception Females must be willing to abide by protocol specified methods to avoid becoming pregnant. Women of childbearing potential must use an adequate form of birth control determined by the investigator (e.g., oral contraceptives, double-barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or vasectomy).
* HIV-1 RNA >1,000 copies/mL at Screening.
* In the opinion of the investigator, subject has a stable CD4+ T lymphocyte count while off ARV and 250 cells/mm3 at Screening.
* Participants should have no clinically significant findings on screening evaluations (clinical, laboratory, or EKG).
* Be able to comprehend and willing to sign an ICF.
* Be able to comply with the protocol requirements.
* Have life expectancy > 6 months.
* Laboratory values obtained during screening must be within normal limits or meet the following requirements (Safety Labs):
* ANC 1000/mm3
* Hemoglobin 9.0 g/dL
* Glucose (nonfasting) <116 mg/dL
* Bilirubin 1.5 x upper limit of normal (ULN)
* Liver function tests (AST & ALT) 1.25 x ULN at screening and baseline
* GGT < 5.0 x ULN
* Negative hepatitis panel obtained less than or equal to 6 months prior to Study Entry
* Creatinine 1.3 x ULN
* Creatine phosphokinase (CPK) 5 x ULN unless further evaluation determines it to be due to exercise
* Urine protein 2+
* Prothrombin time (PT)1.25 x ULN
* Lipase 1.2 x ULN

Exclusion Criteria:

* Current or recent (<3 months) history of opportunistic infection that,
* Acute illness within 1 week of the baseline visit.
* Participant is not able to comply with the dosing schedule and protocol evaluations.
* Participant is anticipated to begin ARV treatment during participation in the study.
* Pregnancy, breastfeeding or postpartum (less than 3 months).
* Diagnosis of diabetes.
* Any condition which could compromise participant safety or adherence to the protocol.
* Documented positive test for hepatitis B surface antigen, hepatitis B surface antibody (with the exception of participants who received hepatitis B vaccination and have hepatitis B surface antibody), hepatitis B core antibody, and hepatitis C antibody.
* Any grade 3 or 4 laboratory abnormality noted at screening according to the DAIDS grading scale (Appendix A), except for the following:
* Grade 3 or 4 triglyceride elevations.
* Grade 3 cholesterol elevation.
* Grade 3 non-fasting glucose elevation.
* Participant has a malabsorption syndrome possibly affecting drug absorption (e.g. Crohn's disease or chronic pancreatitis).
* Participant has received an HIV prophylactic or therapeutic vaccination within 6 months prior to the first dose of study medication.
* Investigational therapy within 30 days prior to the Baseline visit.
* Radiation therapy or systemic cytotoxic chemotherapeutic agents within 12 weeks prior to the baseline visit or have not recovered from side effects from such therapy prior to the first dose of study medication.
* Positive urine screen for drugs of abuse at Screening, unless the investigator deems that the result is associated with a prescribed medication or inhaled use of THC.
* Inability to avoid all tea/tea products (including herbal, caffeinated, decaffeinated, iced tea), apples, chocolate, broad beans (fava beans), plums, prunes, cherries, fruit juices containing apples, cherries, or plums, dietary supplements, and herbal products for 1 week prior to the baseline visit and for the duration of the study.
* Inability to limit caffeine intake to not exceed 12 oz. of caffeinated beverage per day (if espresso, no more than 1 oz. or 1 shot) beginning 2 days prior and for the duration of the study.
* Prior exposure to TNX-355 (an investigational anti-HIV agent that binds to the CD4+ T lymphocyte surface).
* Participant has used proton pump inhibitors starting 14 days before Study Day 1 and is unable to avoid taking proton pump inhibitors for the duration of the study.
* Participant has used H2 blockers starting 24 hours before Study Day 1 and is unable to avoid taking H2 blockers for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Seeborg, MD, MPH, Principal Investigator — Baylor College of Medicine; Roberto Arduino, MD, Study Director — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyphenon E 1600 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Four capsules twice a day.
  Polyphenon E: There will be 3 dose levels and for each dose level, there will be 6 subjects who will receive the study drug and 2 subjects who will be randomized to take placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 2400 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Six capsules twice a day.
  Polyphenon E: There will be 3 dose levels and for each dose level, there will be 6 subjects who will receive the study drug and 2 subjects who will be randomized to take placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 3200 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Eight capsules twice a day.
  Polyphenon E: There will be 3 dose levels and for each dose level, there will be 6 subjects who will receive the study drug and 2 subjects who will be randomized to take placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Placebo: No active drug (Polyphenon E) was administered
Period: Overall Study
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day | Placebo
Started | 6 | 6 | 5 | 6
Completed | 6 | 5 | 5 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Polyphenon E 1600 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Four capsules twice a day.
  Polyphenon E: There will be three treatment arms, each consisting of 6 participants. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 2400 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Six capsules twice a day.
  Polyphenon E: There will be three treatment arms, each consisting of 6 participants. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 3200 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Eight capsules twice a day.
  Polyphenon E: There will be three treatment arms, each consisting of 6 participants. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Placebo: No active drug (Polyphenon E) is given in the Placebo group. A total of 6 participants will be in the Placebo group. 2 participants from the Placebo group will be paired with each of the active treatment groups.
  Safety data from all participants will be evaluated.
- Total: Total of all reporting groups
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 6 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.65 (11.5290) | 28.5166 (6.3857) | 27.3666 (4.6161) | 34.7666 (9.2310) | 31.3249 (3.4079)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 5 | 12
  Male | 5 | 1 | 4 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 4 | 4 | 15
  White | 4 | 1 | 1 | 2 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 5 | 6 | 23
CD4 count [Median (Inter-Quartile Range); unit: cell count (10^6 cells/L)] | 380 [188 to 698] | 594 [188 to 1173] | 432 [408 to 857] | 558.5 [372.3 to 827] | 509 [237 to 985]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety of Polyphenon E (800mg, 1200mg, 1600mg EGCG twice daily for 14 days) in HIV-1-infected subjects.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Polyphenon E 1600 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Four capsules twice a day.
  Polyphenon E: There will be three treatment arms, each consisting of 8 participants. Two participants in each study arm will be randomized to receive placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 2400 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Six capsules twice a day.
  Polyphenon E: There will be three treatment arms, each consisting of 8 participants. Two participants in each study arm will be randomized to receive placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 3200 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Eight capsules twice a day.
  Polyphenon E: There will be three treatment arms, each consisting of 8 participants. Two participants in each study arm will be randomized to receive placebo. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each arm is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6
Participants
  Grade 1 AE Grade 1 AE- Mild; asymptomatic or mild symptoms, intervention not indicated | 1 | 2 | 3 | 0
  Grade 2 AE- Moderate; minimal, local or noninvasive intervention indicated | 0 | 0 | 0 | 0
  Grade 3 AE- Severe; but not immediately life-threatening; hospitalization indicated; disabling | 0 | 0 | 0 | 0
  Grade 4 AE- Life-threatening consequences; urgent intervention indicated. | 0 | 0 | 0 | 0
  Grade 5 AE- Death related to AE | 0 | 0 | 0 | 0

2. Primary Outcome: Median Change of log10 HIV-1 RNA Copies/ml
Description: Median change of log10 HIV-1 RNA copies/ml from baseline in subjects who have completed 14 days of treatment (800mg, 1200mg, 1600mg EGCG bid) or placebo.
Time Frame: Baseline and 14 days
Measure: Median (Inter-Quartile Range); unit: log10 HIV RNA copies/ml
Groups:
- Placebo Placebo: No active drug (Polyphenon E) was administered
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day | Placebo Placebo
Number analyzed (Participants) | 5 | 5 | 4 | 4
log10 HIV RNA copies/ml | 0.01 [-0.13 to 0.80] | -0.07 [-0.18 to 0.58] | 0.17 [-0.05 to 0.20] | 0.01 [-0.18 to 0.07]
Statistical Analysis 1: Comparison: Polyphenon E 1600 mg/Day vs Polyphenon E 2400 mg/Day vs Polyphenon E 3200 mg/Day vs Placebo Placebo; The study hypothesis tested whether Polyphenon E given twice daily for 14 days at the specified doses has an effect on antiviral activity compared with placebo, measured by differences from baseline to day 14 in plasma HIV-1 RNA level (log10 copies/mL). The Wilcoxon signed-rank test was used to test the null hypothesis that there was no change at Day 14 versus baseline; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Polyphenon E 1600 mg/Day vs Polyphenon E 2400 mg/Day vs Polyphenon E 3200 mg/Day vs Placebo Placebo; Test type: Superiority; p = 0.74, Kruskal-Wallis — Analysis was stratified by treatment group. The Kruskal-Wallis test was used to compare the change of log10 HIV-1 RNA copies/ml between treatment groups

3. Secondary Outcome: Number of Participants Achieving > 0.75 or 1.0 log10 Reduction in HIV-1 RNA or <400 Copies/ml
Description: The number of participants achieving >0.75 or 1.0 log10 reduction in HIV-1 RNA or <400 copies/ml with 14 days of Polyphenon E (800mg, 1200mg, or 1600mg EGCG bid) or placebo.
Time Frame: Baseline to 14 days
Measure: Number; unit: participants
Groups:
- Placebo: Placebo
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6
participants | 0 | 0 | 0 | 0

4. Secondary Outcome: The Mean Change in CD4+ T Lymphocyte Counts
Description: The mean change in CD4+ T lymphocyte counts when participants have had Polyphenon E (800mg, 1200mg, 1600mg EGCG bid for 14 days).
Time Frame: Baseline to 14 days
Measure: Mean (Standard Deviation); unit: 10^6 cells/L
Groups:
- Placebo Placebo: Placebo
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day | Placebo Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6
10^6 cells/L | 11.833333 (14.282857) | 16.166667 (14.282857) | 11.800000 (13.416408) | 8.166667 (14.282857)

5. Secondary Outcome: Composite of Pharmacokinetics Time Frame: Predose, 0,0.5,1,1.5,2,3,4,6,8,12 Hours Post-dose
Description: Plasma PK parameters of EGCG after single dose and at steady state (after 14 day EGCG treatment).
Time Frame: Predose, 0,0.5,1,1.5,2,3,4,6,8,12 Hours Post-dose on Days 1 and 14
Population: The number of subjects who received treatment with Polyphenon E in each arm for each pharmacokinetic outcome measure [t1/2 (h), Cmax (ng/ml), AUC 0-12h (h*ng/ml), CL/F (L/h). Day14:Day1 ratio reported as geometric mean (90% confidence interval).
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day
Number analyzed (Participants) | 6 | 5 | 5
Ratio
  t 1/2 | 1.08 [0.74 to 1.56] | 1.14 [0.9 to 1.43] | 0.9 [0.69 to 1.18]
  Cmax | 1.21 [0.78 to 1.9] | 1.33 [0.65 to 2.74] | 0.65 [0.45 to 0.92]
  AUC 0-12 | 1.4 [1.08 to 1.82] | 1.28 [0.61 to 2.69] | 0.88 [0.63 to 1.22]
  CL/F | 0.75 [0.58 to 0.97] | 0.81 [0.4 to 1.67] | 1.21 [0.86 to 1.71]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the 14-day study period and 7- day follow up period for a total of 21 days
Groups:
- Polyphenon E 1600 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Four capsules twice a day.
  Polyphenon E: There will be three dose levels, each consisting of 6 participants. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding arm will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each dose level is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each dose level. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 2400 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Six capsules twice a day.
  Polyphenon E: There will be three dose levels, each consisting of 6 participants. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding dose level will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each dose level is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Polyphenon E 3200 mg/Day: Drug: Polyphenon E Polyphenon E capsules containing 200 mg of epigallocatechin-gallate. Eight capsules twice a day.
  Polyphenon E: There will be three dose levels, each consisting of 6 participants. Dosing will be escalated sequentially contingent on the safety profile of previous doses. Safety data from all participants receiving Polyphenon® E in the preceding dose level will be evaluated and considered acceptable prior to escalation to the next higher dose. PK analyses will be also performed as each dose level is completed. It is necessary to confirm EGCG pharmacokinetics in the event that the primary outcome measure of virologic response is not observed for each arm. For each PK visit on Study Days 1 and 14, a total of 10 blood samples will be obtained per subject.
- Placebo: No active drug (Polyphenon E) is given in the Placebo group. A total of 6 subjects will be in the placebo group. 2 subjects will be randomized to take placebo in each of the active treatment groups.
  Safety data from all participants will be evaluated.
Arm/Group | Polyphenon E 1600 mg/Day | Polyphenon E 2400 mg/Day | Polyphenon E 3200 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 3/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyphenon E 1600 mg/Day (N=6) | Polyphenon E 2400 mg/Day (N=6) | Polyphenon E 3200 mg/Day (N=5) | Placebo (N=6)
Mild abdominal cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased carbon dioxide (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated lipase (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated SGPT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased serum calcium (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated SGOT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated serum protein (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased serum Magnesium level (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes